CLINICAL TRIAL: NCT06088017
Title: A Phase I Clinical Trial to Compare and Evaluate the Safety and Pharmacokinetic Characteristics After Administration of CKD-391(2) and Co-administration of CKD-331 and D337 in Healthy Adult Volunteers
Brief Title: A Clinical Trial to Compare and Evaluate the Safety and Pharmacokinetics of CKD-391(2)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A52_11BE2309
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2023-10

CONDITIONS: Dyslipidemias
Keywords: CKD-391; CKD-391(2)
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): * Period 1: CKD-331, D337 - A single oral dose of 2 tablets under fasting condition
  * Period 2: CKD-391(2) - A single oral dose of 1 tablet under fasting condition
  * Period 3: CKD-331, D337 - A single oral dose of 2 tablets under fasting condition
  * Period 4: CKD-391(2) - A single oral dose of 1 tablet under fasting condition
  Interventions: Drug: CKD-391(2); Drug: CKD-331, D337
- Sequence 2 (Experimental): * Period 1: CKD-391(2) - A single oral dose of 1 tablet under fasting condition
  * Period 2: CKD-331, D337 - A single oral dose of 2 tablets under fasting condition
  * Period 3: CKD-391(2) - A single oral dose of 1 tablet under fasting condition
  * Period 4: CKD-331, D337 - A single oral dose of 2 tablets under fasting condition
  Interventions: Drug: CKD-391(2); Drug: CKD-331, D337

INTERVENTIONS:
Drug: CKD-391(2) — QD, PO
Drug: CKD-331, D337 — QD, PO

SUMMARY:
A clinical trial to compare and evaluate the safety and pharmacokinetics of CKD-391(2)

DETAILED DESCRIPTION:
A phase I clinical trial to compare and evaluate the safety and pharmacokinetic characteristics after administration of CKD-391(2) and co-administration of CKD-331 and D337 in healthy adult volunteers

ELIGIBILITY:
* Inclusion Criteria

  1. Healthy adult aged between 19 to 55 at screening
  2. Weight ≥ 50kg(man) or 45kg(woman), with calculated body mass index (BMI) of 18 to 30kg/m2
  3. Those who have no clinically significant congenital or chronic diseases and have no abnormal symptoms of findings
  4. Those who are deemed suitable for clinical trials based on laboratory (hematology, blood chemistry, serology, urinalysis, urine drug test) and 12-lead ECG results at screening
  5. Those who agree to contraception from the first IP dosing day till 14 days after the last dosing day and decide not to provide sperm during the participation of clinical trial
  6. Those who voluntarily decide to participate in paper and agree to comply with the cautions after fully understand the detailed description of this clinical trial
* Exclusion Criteria

  1. Those who have used drugs that induce or inhibit drug metabolizing enzymes, such as barbiturates, within 1 month before the first dosing date, or who have used drugs that may interfere with this study within 10 days before the first dosing day
  2. Those who exceed an alcohol, caffeine and cigarette consumption (caffeine> 5 cups/day, alcohol> 21 glasses/week(man), 14 glasses/week(woman), smoking> 20 cigarettes/day) and not able to stop on smoking, caffeine and alcohol
  3. Those who received investigational products or participated in bioequivalence test within 6 months before the first administration of clinical trial drugs
  4. Those who donated whole blood within 8 weeks before the first date of administration and donated ingredients within 2 weeks or received blood transfusion in 4 weeks
  5. Those who have a history of gastrointestinal surgery except simple appendectomy and hernia surgery
  6. Patients with the following diseases
* Patients with active liver disease or with elevated amino transferase levels with unknown cause increased by more than 3 times the normal upper limit
* Patients with severe liver failure or biliary obstruction and bile congestion
* Patients with muscular disease, rhabdomyolysis, or persons with a past history
* Patients with hypothyroidism, patients with genetic muscle disease or their family history, and patients with history of muscle disability due to drugs
* Patients with renal impairment or a history of in and patients with severe renal dysfunction
* Patients with a history of muscle toxicity to other statin drugs or fibrate drugs

  7. Those who have genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption

  8. Those who have hypersensitivity to the main constituents or components of the investigational drug

  9. Those who have a history of drug abuse within 1 year of screening or who have tested positive for urine drug tests

  10. Woman who are pregnant or breastfeeding

  11. Those who are deemed insufficient to participate in clinical study by investigators

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-01-07 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
AUCt of CKD-391(2) | Pre-dose(0 hour) to 72hours
  Area under the concentration-time curve time zero to time
Cmax of CKD-391(2) | Pre-dose(0 hour) to 72hours
  Maximum plasma concentration of the drug

CONTACTS AND LOCATIONS:
Locations (1):
- Bumin hopspital, Seoul, Seoul, Gangseo-gu, South Korea

IPD SHARING:
Plan to Share IPD: No